CLINICAL TRIAL: NCT06939868
Title: Effectiveness of 'Cepham Supplement' on Hot Flash Severity/Frequency and Menopausal Symptoms in Postmenopausal Women: A Randomized Double-Blind Placebo-Controlled Trial
Brief Title: Effect of a Cepham Supplement on Hot Flashes and Menopausal Symptoms in Postmenopausal Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jacksonville University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SterlingIRB2025
Record Dates: First submitted 2025-04-11; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: D008593
Keywords: menopause; hot flashes; supplement
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplement Group (Active Comparator)
  Interventions: Dietary Supplement: Shatavari Root Extract, oral capsule
- Placebo Group: Sugar pill (Placebo Comparator)
  Interventions: Dietary Supplement: Shatavari Root Extract, oral capsule

INTERVENTIONS:
Dietary Supplement: Shatavari Root Extract, oral capsule — This intervention consists of a proprietary, standardized extract of Asparagus racemosus (Shatavari), formulated specifically for women's health and cognitive support. The supplement is provided in oral capsule form and standardized to a specific concentration of shatavarin IV, the primary active compound. Participants will take one capsule daily for 30 days.
  This formulation, known as SheVari4™, is patent-pending and manufactured by Cepham, designed to address vasomotor symptoms (hot flashes) and other menopausal concerns. It is distinct from other Shatavari supplements in its standardization and use in a placebo-controlled, double-blind trial targeting postmenopausal women.

SUMMARY:
The goal of this clinical trial is to learn if a daily nutritional supplement can reduce hot flashes and other menopausal symptoms in postmenopausal women.

The main questions this study aims to answer are:

Does the supplement reduce the number and severity of daily hot flashes?

Does it improve other common menopausal symptoms?

Researchers will compare the supplement to a placebo (a look-alike capsule with no active ingredients) to see if it helps manage symptoms during menopause.

Participants will:

Take either the supplement or a placebo daily for 30 days

Track their hot flashes each day using a short online survey

Complete a symptom questionnaire at the beginning and end of the study

This study is for women ages 40-60 who have been postmenopausal for at least one year and currently experience bothersome hot flashes.

DETAILED DESCRIPTION:
Purpose:

To evaluate the effectiveness of a nutritional supplement in reducing hot flash severity/frequency and menopausal symptoms in postmenopausal women.

Design:

Randomized, double-blind, placebo-controlled, two-arm, parallel-group trial over 30 days.

Participants:

Women aged 40-60 who are postmenopausal (≥1 year without menses) and report bothersome hot flashes (Menopause Rating Scale score ≥14, and hot flash severity of 3 or 4).

Exclusion Criteria:

Current hormone therapy or medications affecting hot flashes; significant comorbidities.

Intervention:

Group 1: Placebo

Group 2: Supplement

Assessments:

Daily self-reports of hot flash frequency/severity

Menopausal symptom assessments at baseline (Day 0) and post-intervention (Day 30)

Outcomes:

Primary: Hot flash severity and frequency

Secondary: Overall menopausal symptoms

ELIGIBILITY:
Inclusion Criteria:

* Adult women aged 40-60 years.
* Menopause Rating Scale score: (a) GE 14 and (b) score of 3 or 4 (severe to very severe) for hot flashes (Blumel et al., 2018).

Exclusion Criteria:

* Current use of hormone therapy or other medications known to affect hot flashes.
* Significant comorbidities that may interfere with study participation.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 44 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Composite hot flash score: Frequency × Severity | 30 days
  Frequency: Total number of hot flashes experienced that day. Hot Flash Severity: Rating of hot flashes on a 7-point severity scale (0 = none, 1 = very mild, 2 = mild, 3 = mild/moderate, 4 = moderate, 5 = severe, 6 = very severe)

SECONDARY OUTCOMES:
Menopause Rating Scale | 30 days
  Validated self-administered questionnaire consisting of 11 items that assesses menopausal symptoms. Each item is rated on a 5-point Likert scale from 0 (not present) to 4 (very severe), yielding a total score range of 0 to 44, with higher scores indicating more severe symptoms. The Menopause Rating Scale is divided into three domains: somatic (hot flashes, heart discomfort, sleep problems, joint and muscular discomfort), psychological (depressive mood, irritability, anxiety, physical and mental exhaustion), and urogenital (sexual problems, bladder problems, vaginal dryness). This scale has been widely used in clinical research to quantify menopausal symptom burden and its impact on quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Heather A Hausenblas, PhD, Principal Investigator — Jacksonville University
Locations (1):
- Jacksonville University, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No